CLINICAL TRIAL: NCT04344600
Title: Peginterferon Lambda-1a for the Prevention and Treatment of SARS-CoV-2 Infection
Brief Title: Peginterferon Lambda-1a for the Prevention and Treatment of SARS-CoV-2 (COVID-19) Infection
Acronym: PROTECT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Single center study with low enrollment
Sponsor: Johns Hopkins University (Other)
Collaborators: Eiger BioPharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00248163
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Results first posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Sars-CoV-2 Infection
Keywords: SARS-CoV-2; COVID-19; Lambda interferon
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, single-blind, controlled trial
Who Masked: Participant
Masking Description: Single-blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Peginterferon lambda alfa-1a (Experimental): peginterferon lambda-1a (Lambda) 180 micrograms by subcutaneous injection for participants who are not infected with SARS-CoV-2
  Interventions: Drug: Peginterferon lambda alfa-1a subcutaneous injection
- Placebo (Placebo Comparator): Placebo (saline) by subcutaneous injection for participants who are not infected with SARS-CoV-2
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Peginterferon lambda alfa-1a subcutaneous injection — Peginterferon lambda-1a 180 micrograms by subcutaneous injection
  Arms: Peginterferon lambda alfa-1a
Other: Saline — Saline subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a phase 2b prospective, randomized, single-blind, controlled trial of a single subcutaneous injection of peginterferon lambda-1a versus placebo for prevention of SARS-CoV-2 infection in non-hospitalized participants at high risk for infection due to household exposure to an individual with coronavirus disease (COVID-19). The study will also evaluate the regimens participants with asymptomatic SARS-CoV-2 infection detected at study entry. All participants will be followed for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Peripheral capillary oxygen saturation (SpO2) ≥ 95% on room air at screening
* Age ≥18 years

Exclusion Criteria:

* Hospitalized or impending hospitalization at the time of screening
* Symptoms of cough, fever or shortness of breath within 72 hours
* Prior or current treatment with other experimental or approved agents targeting SARS-CoV-2 or SARS-CoV-1
* Positive pregnancy test
* Active autoimmune disease or sarcoidosis (with the exception of controlled thyroid disease)
* Active decompensated liver disease (ascites, encephalopathy)
* Active congestive heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sulkowski, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hemann EA, Gale M Jr, Savan R. Interferon Lambda Genetics and Biology in Regulation of Viral Control. Front Immunol. 2017 Dec 6;8:1707. doi: 10.3389/fimmu.2017.01707. eCollection 2017. PMID 29270173
- [Background] Mordstein M, Neugebauer E, Ditt V, Jessen B, Rieger T, Falcone V, Sorgeloos F, Ehl S, Mayer D, Kochs G, Schwemmle M, Gunther S, Drosten C, Michiels T, Staeheli P. Lambda interferon renders epithelial cells of the respiratory and gastrointestinal tracts resistant to viral infections. J Virol. 2010 Jun;84(11):5670-7. doi: 10.1128/JVI.00272-10. Epub 2010 Mar 24. PMID 20335250
- [Background] Loutfy MR, Blatt LM, Siminovitch KA, Ward S, Wolff B, Lho H, Pham DH, Deif H, LaMere EA, Chang M, Kain KC, Farcas GA, Ferguson P, Latchford M, Levy G, Dennis JW, Lai EK, Fish EN. Interferon alfacon-1 plus corticosteroids in severe acute respiratory syndrome: a preliminary study. JAMA. 2003 Dec 24;290(24):3222-8. doi: 10.1001/jama.290.24.3222. PMID 14693875
- [Derived] Lee JS, Shin EC. The type I interferon response in COVID-19: implications for treatment. Nat Rev Immunol. 2020 Oct;20(10):585-586. doi: 10.1038/s41577-020-00429-3. PMID 32788708
- See also: WHO COVID-19 landscape analysis of therapeutics. — https://www.who.int/blueprint/priority-diseases/key-action/novel-coronavirus/en/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peginterferon Lambda Alfa-1a | Placebo
Started | 2 | 4
Completed | 2 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginterferon Lambda Alfa-1a | Placebo | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With no Evidence of SARS-CoV-2 Infection
Description: Number of participants with no evidence of SARS-CoV-2 infection at or before study day 28.
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Peginterferon Lambda Alfa-1a | Placebo
Number analyzed (Participants) | 2 | 4
Participants | 2 | 4

2. Secondary Outcome: Time to no Detection of SARS-CoV-2
Description: Resolution of SARS-CoV-2 infection in the upper respiratory tract as assessed by time (in days) to no detection of SARS-CoV-2 in two upper respiratory samples.
Time Frame: Up to 14 days
Population: This outcome was not assessed because all participants were negative at the time of entering study and didn't test positive. No data was collected.
Arm/Group | Peginterferon Lambda Alfa-1a | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of informed consent through protocol Day 28
Arm/Group | Peginterferon Lambda Alfa-1a | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 0/2 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT04344600/Prot_SAP_002.pdf